CLINICAL TRIAL: NCT06495281
Title: A Observational Study to Evaluate Effectiveness, Safety of Triple Combination Therapy of Zemidapa and Metformin in Patients With Type 2 DM Who Received Double or Triple Combination Therapy Including DPP4-inhibitor Other Than Gemigliptin
Brief Title: Observational Study of Triple Combination Therapy of Zemidapa Tab. and Metformin in Type 2 Diabetes Mellitus Patients
Status: Recruiting | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-GLOS001
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of the triple combination therapy of Zemidapa Tab. and Metformin in patients with type 2 diabete mellitus

ELIGIBILITY:
Inclusion Criteria:

* type 2 DM Patients who are receiving one of the following three therapies during which the patients are prescribed with Zemidapa Tab. for the first time at the discretion of the attending physician:

  1. Double combination therapy (Metformin and a DPP-4 inhibitor other than Gemigliptin)
  2. Triple combination therapy (Metformin, a DPP-4 inhibitor other than Gemigliptin, and a SGLT-2 inhibitor)
  3. Triple combination therapy (Metformin, a DPP-4 inhibitor other than Gemigliptin, and Sulfonylurea [SU])
* patients with HbA1c results and who signed the written consent form

Exclusion Criteria:

- Patients contraindicated for the approved use of Zemidapa Tab. or have participated in another clinical study within 12 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, secondary and tetiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline of HbA1c at 12 weeks | baseline, 12 weeks

SECONDARY OUTCOMES:
the rate of subjects who reached the target value of less than 7% HbA1c | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea